CLINICAL TRIAL: NCT04412538
Title: A Randomized, Double-blind, Placebo-controlled, Phase Ia/IIa Trial of an Inactivated SARS-CoV-2 Vaccine in Healthy People Aged 18 to 59 Years
Brief Title: Safety and Immunogenicity Study of an Inactivated SARS-CoV-2 Vaccine for Preventing Against COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: West China Second University Hospital (Other); Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20200401
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Low dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of low dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- Low dosage vaccine on a 0- and 14-day schedule (Experimental): Two doses of low dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 14
  Interventions: Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule
- Medium dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of medium dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- Medium dosage vaccine on a 0- and 14-day schedule (Experimental): Two doses of medium dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 14
  Interventions: Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule
- High dosage vaccine on a 0- and 28-day schedule (Experimental): Two doses of high dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 28
  Interventions: Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule
- High dosage vaccine on a 0- and 14-day schedule (Experimental): Two doses of high dosage Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0, 14
  Interventions: Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule
- Placebo on a 0- and 28-day schedule (Placebo Comparator): Two doses of placebo at the vaccination schedule of day 0, 28
  Interventions: Biological: Placebo on a 0- and 28-day schedule
- Placebo on a 0- and 14-day schedule (Placebo Comparator): Two doses of placebo at the vaccination schedule of day 0, 14
  Interventions: Biological: Placebo on a 0- and 14-day schedule

INTERVENTIONS:
Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of low dosage(50U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: Low dosage vaccine on a 0- and 28-day schedule
Biological: Low dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule — Two doses of low dosage(50U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,14
  Arms: Low dosage vaccine on a 0- and 14-day schedule
Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of medium dosage(100U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: Medium dosage vaccine on a 0- and 28-day schedule
Biological: Medium dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule — Two doses of medium dosage(100U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,14
  Arms: Medium dosage vaccine on a 0- and 14-day schedule
Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 28-day schedule — Two doses of high dosage(150U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,28
  Arms: High dosage vaccine on a 0- and 28-day schedule
Biological: High dosage Inactivated SARS-CoV-2 Vaccine on a 0- and 14-day schedule — Two doses of high dosage(150U/0.5ml) Inactivated SARS-CoV-2 Vaccine at the vaccination schedule of day 0,14
  Arms: High dosage vaccine on a 0- and 14-day schedule
Biological: Placebo on a 0- and 28-day schedule — Two doses of placebo at the vaccination schedule of day 0,28
  Arms: Placebo on a 0- and 28-day schedule
Biological: Placebo on a 0- and 14-day schedule — Two doses of placebo at the vaccination schedule of day 0,14
  Arms: Placebo on a 0- and 14-day schedule

SUMMARY:
This study is a randomized, double-blinded, and placebo-controlled phase Ia/IIa clinical trial of the Inactivated SARS-CoV-2 Vaccine to evaluate the safety and immunogenicity of the vaccine in healthy people aged 18~59 Years.

DETAILED DESCRIPTION:
This phase Ia/IIa trial is designed to evaluate the safety and immunogenicity of different doses of the Inactivated SARS-CoV-2 Vaccine inoculated with different immunization schedules based upon the randomized, double-blind and placebo-controlled principle. A total of 942 subjects aged 18 to 59 years old will be enrolled in the study, of which 192 and 750 will be enrolled for phase Ia and phase Ⅱa,respectively.The enrolled subjects in phase Ia receive two doses of low-, medium-, or high-dose of experimental vaccines or placebo at an interval of 14 or 28 days, while the enrolled subjects in Phase Ⅱa receive two doses of medium, high-dose experimental vaccines or placebo at an interval of 14 or 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Phase Ia:

  1. Healthy adults aged 18 to 59 years (including boundary values), both men and women.
  2. Proven legal identity.
  3. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
  4. Participants should be able to communicate well with investigators, understand and comply with the requirements of this trial.
  5. Axillary temperature ≤37.0 ℃.
* Phase IIa:

  1. Healthy adults aged 18 to 59 years (including boundary values), both men and women.
  2. Proven legal identity.
  3. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
  4. Participants should be able to communicate well with investigators, understand and comply with the requirements of this trial.
  5. Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Phase Ia:

  1. Contraindications for vaccination.
  2. History of allergy to vaccines or drugs.
  3. Immunization with any vaccine within 1 month.
  4. History of abnormal clinical manifestations and serious diseases to be excluded, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other system diseases, and a history of malignant tumors.
  5. Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
  6. Those who have a hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis or bleeding disorders.
  7. Those who cannot tolerate venipuncture, or have a history of halo needles or halo blood.
  8. Surgical removal of spleen or other important organs for any reason.
  9. Those who have undergone surgery within 3 months before signing the informed consent, or those who plan to perform surgery during the trial or within 3 months after the end of the trial (including cosmetic surgery, dental and oral surgery).
  10. Those who donated or lost blood (≥400 mL) in the past 3 months, who received blood transfusion or use of blood products, or who planned blood donation during the trial.
  11. Receipt of other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months, or plan to use other investigational or unregistered products during the study.
  12. Receipt of immunosuppressive therapy within 6 months before signing the informed consent form, such as long-term systemic glucocorticoid therapy (with systemic glucocorticoid therapy for more than 2 weeks within 6 months, such as prednisone or similar drugs) ), but local administration (such as ointment, eye drops, inhalation, or nasal spray) is allowed. The local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure.
  13. Those who have took soft drugs (such as marijuana) within 3 months before signing the informed consent form or took hard drugs (such as: cocaine, phencyclidine, etc.) within 1 year before the trial.
  14. Those who smoked more than 5 cigarettes per day within 3 months before signing the informed consent form.
  15. The weekly drinking volume is greater than 14 units within 3 months before signing the informed consent form (1 unit alcohol approximately equal to 360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine).
  16. The comprehensive physical examination does not meet the health standards, mainly including: (1) Those with abnormal vital signs with clinical significance. (2) BMI<18 kg/m^2 or> 30 kg/m^2. (3) Abnormal laboratory examination with clinical significance. (4) Those who tested positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B e antigen, hepatitis C virus antibody, or Treponema pallidum antibody (tp-trust).
  17. Participants who have a positive pregnancy test, or are breastfeeding, or plan to become pregnant, or plan to donate sperm or eggs from the screening to 12 months after the second vaccination.
  18. Positive in drug abuse screening during the screening period (Morphine, Methamphetamine, Ketamine, MDMA and Tetrahydrocannabinolic acid).
  19. Positive in alcohol breath test during the screening period.
  20. Positive in SARS-CoV-2 nucleic acid screening or antibodies (IgG or IgM) screening.
  21. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or other coronavirus infection (HCoV-229E, HCoV-OC43, HCoV-NL63, HCoV-HKU1).
  22. History of contact with confirmed or suspected cases infected with SARS-CoV-2 within 1 month.
  23. Any other situations judged by investigators as not suitable for participating in this study.
* Phase IIa:

  1. Contraindications for vaccination.
  2. History of allergy to vaccines or drugs.
  3. Immunization with any vaccine within 1 month.
  4. History of abnormal clinical manifestations and serious diseases to be excluded, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other system diseases, and a history of malignant tumors.
  5. Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
  6. Those who have a hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis or bleeding disorders.
  7. Surgical removal of spleen or other important organs for any reason.
  8. Those who have undergone surgery within 3 months before signing the informed consent, or those who plan to perform surgery during the trial or within 3 months after the end of the trial (including cosmetic surgery, dental and oral surgery).
  9. Those who donated or lost blood (≥400 mL) in the past 3 months, who received blood transfusion or use of blood products, or who planned blood donation during the trial.
  10. Receipt of other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months, or plan to use other investigational or unregistered products during the study.
  11. Receipt of immunosuppressive therapy within 6 months before signing the informed consent form, such as long-term systemic glucocorticoid therapy (with systemic glucocorticoid therapy for more than 2 weeks within 6 months, such as prednisone or similar drugs) ), but local administration (such as ointment, eye drops, inhalation, or nasal spray) is allowed. The local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure.
  12. The comprehensive physical examination does not meet the health standards, mainly including: (1) Those with abnormal vital signs (Pulse <55 beats per minute or> 100 beats per minute at rest, Systolic blood pressure ≥140mmHg or Diastolic blood pressure ≥90mmHg, breathing> 20 beats per minute or <12 beats per minute). (2) Those who tested positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B e antigen, hepatitis C virus antibody, or Treponema pallidum antibody (tp-trust).
  13. Participants who have a positive pregnancy test, or are breastfeeding, or plan to become pregnant, or plan to donate sperm or eggs from the screening to 12 months after the second vaccination.
  14. Positive in SARS-CoV-2 nucleic acid screening or antibodies (IgG or IgM) screening.
  15. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or other coronavirus infection (HCoV-229E, HCoV-OC43, HCoV-NL63, HCoV-HKU1).
  16. History of contact with confirmed or suspected cases infected with SARS-CoV-2 within 1 month.
  17. Any other situations judged by investigators as not suitable for participating in this study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 942 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse reactions/events rate | 7 days after vaccination
  Occurence of adverse reactions/events after vaccination
Adverse reactions/events rate | 28 days after vaccination
  Occurence of adverse reactions/events after vaccination
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase IIa (Day 0, 14 schedule) | 14 days after the second vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for the Phase IIa immunization schedule of day 0,14
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for the Phase IIa immunization schedule of day 0,28
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase IIa (Day 0, 14 schedule) | 14 days after the second vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,14
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,28

SECONDARY OUTCOMES:
Serious adverse events | 12 months after the second vaccination
  Occurence of Serious adverse events after vaccination
Level of Neutralizing antibodies against SARS-CoV-2 Phase Ia (Day 0, 14 schedule) | 7, 14 and 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for the Phase Ia immunization schedule of day 0,14
Level of Neutralizing antibodies against SARS-CoV-2 Phase IIa (Day 0, 14 schedule) | 14 and 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for the Phase IIa immunization schedule of day 0,14
Level of IgG antibodies against SARS-CoV-2 Phase Ia (Day 0, 14 schedule) | 7, 14 and 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,14
Level of IgG antibodies against SARS-CoV-2 Phase IIa (Day 0, 14 schedule) | 14 and 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,14
Level of Neutralizing antibodies against SARS-CoV-2 Phase Ia (Day 0, 28 schedule) | 7 and 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for the Phase Ia immunization schedule of day 0,28
Level of Neutralizing antibodies against SARS-CoV-2 Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for the Phase IIa immunization schedule of day 0,28
Level of IgG antibodies against SARS-CoV-2 Phase Ia (Day 0, 28 schedule) | 7 and 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,28
Level of IgG antibodies against SARS-CoV-2 Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,28
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase Ia (Day 0, 14 schedule) | 14 days after the second vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for the Phase Ia immunization schedule of day 0,14
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase Ia (Day 0, 14 schedule) | 14 days after the second vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,14
Seroconversion rate of Neutralizing antibodies against SARS-CoV-2 Phase Ia (Day 0, 28 schedule) | 28 days after the second vaccination
  Seroconversion rate of neutralizing antibodies against SARS-CoV-2 in serum for the Phase Ia immunization schedule of day 0,28
Seroconversion rate of IgG antibodies against SARS-CoV-2 Phase Ia (Day 0, 28 schedule) | 28 days after the second vaccination
  Seroconversion rate of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,28

OTHER OUTCOMES:
Level of IgM antibodies against SARS-CoV-2 Phase Ia (Day 0, 14 schedule) | 7, 14 and 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,14
Level of IgM antibodies against SARS-CoV-2 Phase IIa (Day 0, 14 schedule) | 14 and 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,14
Level of anti-N protein antibodies Phase Ia (Day 0, 14 schedule) | 7, 14 and 28 days after the second vaccination
  Level of anti-N protein antibodies for the Phase Ia immunization schedule of day 0,14
Level of anti-N protein antibodies Phase IIa (Day 0, 14 schedule) | 14 and 28 days after the second vaccination
  Level of anti-N protein antibodies for the Phase IIa immunization schedule of day 0,14
Level of IgM antibodies against SARS-CoV-2 Phase Ia (Day 0, 28 schedule) | 7 and 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase Ia immunization schedule of day 0,28
Level of IgM antibodies against SARS-CoV-2 Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Level of IgM antibodies against SARS-CoV-2 tested by ELISA in serum for the Phase IIa immunization schedule of day 0,28
Level of anti-N protein antibodies Phase Ia (Day 0, 28 schedule) | 7 and 28 days after the second vaccination
  Level of anti-N protein antibodies for the Phase Ia immunization schedule of day 0,28
Level of anti-N protein antibodies Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Level of anti-N protein antibodies for the Phase IIa immunization schedule of day 0,28
Level of Neutralizing antibodies against SARS-CoV-2 Phase Ia (both schedules) | 3, 6, 9 and 12 months after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for both the Phase Ia immunization schedules
Level of Neutralizing antibodies against SARS-CoV-2 Phase IIa (both schedules) | 6 and 12 months after the second vaccination
  Level of neutralizing antibodies against SARS-CoV-2 in serum for both the Phase IIa immunization schedules
Level of IgG antibodies against SARS-CoV-2 Phase Ia (both schedules) | 3, 6, 9 and 12 months after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for both the Phase Ia immunization schedules
Level of IgG antibodies against SARS-CoV-2 Phase IIa (both schedules) | 6 and 12 months after the second vaccination
  Level of IgG antibodies against SARS-CoV-2 tested by ELISA in serum for both the Phase IIa immunization schedules
Cellular immune responses Phase Ia (Day 0, 14 schedule) | 7, 14 and 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for the Phase Ia immunization schedule of day 0,14
Cellular immune responses Phase IIa (Day 0, 14 schedule) | 14 and 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for the Phase IIa immunization schedule of day 0,14
Cellular immune responses Phase Ia (Day 0, 28 schedule) | 7 and 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for the Phase Ia immunization schedule of day 0,28
Cellular immune responses Phase IIa (Day 0, 28 schedule) | 28 days after the second vaccination
  Cellular immune responses (CD4+, CD8+, Th1, Th2, IFN-γ, TNFα, IL-2, IL-6) will be measured for the Phase IIa immunization schedule of day 0,28

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Principal Investigator — West China Second University Hospital; Xiaoqiang Liu, Principal Investigator — Yunnan Center for Disease Control and Prevention
Locations (1):
- West China Second University Hospital, Sichuan University / West China women's and children's Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Pu J, Yu Q, Yin Z, Zhang Y, Li X, Yin Q, Chen H, Long R, Zhao Z, Mou T, Zhao H, Feng S, Xie Z, Wang L, He Z, Liao Y, Fan S, Jiang R, Wang J, Zhang L, Li J, Zheng H, Cui P, Jiang G, Guo L, Xu M, Yang H, Lu S, Wang X, Gao Y, Xu X, Cai L, Zhou J, Yu L, Chen Z, Hong C, Du D, Zhao H, Li Y, Ma K, Ma Y, Liu D, Yao S, Li C, Che Y, Liu L, Li Q. The safety and immunogenicity of an inactivated SARS-CoV-2 vaccine in Chinese adults aged 18-59 years: A phase I randomized, double-blinded, controlled trial. Vaccine. 2021 May 12;39(20):2746-2754. doi: 10.1016/j.vaccine.2021.04.006. Epub 2021 Apr 9. PMID 33875266
- [Derived] Che Y, Liu X, Pu Y, Zhou M, Zhao Z, Jiang R, Yin Z, Xu M, Yin Q, Wang J, Pu J, Zhao H, Zhang Y, Wang L, Jiang Y, Lei J, Zheng Y, Liao Y, Long R, Yu L, Cui P, Yang H, Zhang Y, Li J, Chen W, He Z, Ma K, Hong C, Li D, Jiang G, Liu D, Xu X, Fan S, Cheng C, Zhao H, Yang J, Li Y, Zou Y, Zhu Y, Zhou Y, Guo Y, Yang T, Chen H, Xie Z, Li C, Li Q. Randomized, Double-Blinded, Placebo-Controlled Phase 2 Trial of an Inactivated Severe Acute Respiratory Syndrome Coronavirus 2 Vaccine in Healthy Adults. Clin Infect Dis. 2021 Dec 6;73(11):e3949-e3955. doi: 10.1093/cid/ciaa1703. PMID 33165503